CLINICAL TRIAL: NCT04460456
Title: A Phase 1/1B, Open-Label, Dose Escalation and Expansion Study of SBT6050 Alone and in Combination With PD-1 Inhibitors in Subjects With Advanced Solid Tumors Expressing HER2
Brief Title: A Study of SBT6050 Alone and in Combination With PD-1 Inhibitors in Subjects With Advanced HER2 Expressing Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Silverback Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBT6050-101
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: HER2 Positive Solid Tumors
Keywords: HER2; ERBB2; Immunotherapy; Gastric Cancer; Gastroesophageal junction; Breast Cancer; Triple Negative Breast Cancer; Stomach Cancer; Colorectal Cancer; Gastrointestinal Cancer; Non-Small Cell Lung Cancer; Monoclonal antibody; TLR8; TLR8 agonist; Antibody drug conjugate; Biliary tract cancer; Head and neck cancer; Urothelial cancer; Endometrial cancer; Pembrolizumab; Anti-PD-1 mAb; Cemiplimab
MeSH Terms: conditions — Stomach Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms; Carcinoma, Non-Small-Cell Lung; Biliary Tract Neoplasms; Head and Neck Neoplasms; Endometrial Neoplasms | interventions — pembrolizumab; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SBT6050 Monotherapy (Experimental): Escalating doses of SBT6050 in Part 1 followed by expansion in Part 2 at the recommended dose determined in Part 1.
  Interventions: Drug: SBT6050
- SBT6050 and pembrolizumab (Experimental): Escalating doses of SBT6050 in combination with pembrolizumab in Part 3 followed by expansion in Part 4 at the recommended dose determined in Part 3.
  Interventions: Drug: SBT6050; Drug: pembrolizumab
- SBT6050 and cemiplimab (Experimental): SBT6050 in combination with cemiplimab in Part 5 at the recommended dose determined in Parts 1 and 3.
  Interventions: Drug: SBT6050; Drug: Cemiplimab

INTERVENTIONS:
Drug: SBT6050 — Escalating doses of SBT6050 in Part 1 and recommended dose in Part 2
Drug: pembrolizumab — 400 mg IV
  Arms: SBT6050 and pembrolizumab
Drug: Cemiplimab — 350 mg IV
  Arms: SBT6050 and cemiplimab

SUMMARY:
A first-in-human (FIH) study using SBT6050 and SBT6050 in combination with PD-1 inhibitors in HER2 expressing or amplified advanced malignancies

DETAILED DESCRIPTION:
This study has 5 parts. Part 1 will evaluate the safety, tolerability, and activity of escalating doses of SBT6050 to estimate the maximum tolerated dose (MTD) and determine the dose recommended for Part 2. Part 2 of the study will further evaluate SBT6050 in select HER2 expressing or amplified advanced malignancies.

Part 3 will evaluate the safety, tolerability, and activity of escalating doses of SBT6050 in combination with pembrolizumab to estimate the MTD and determine the dose recommended for Part 4. Part 4 of the study will further evaluate SBT6050 in combination with pembrolizumab in select HER2 expressing or amplified advanced malignancies.

Part 5 of the study will evaluate the safety, tolerability, and activity of SBT6050 in combination with cemiplimab in select HER2 expressing or amplified advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic HER2-expressing (IHC 2+ or 3+) or amplified solid tumor
* Subjects must have received prior therapies known to confer clinical benefit (unless ineligible or refused to receive)
* Measurable disease per RECIST 1.1
* Tumor lesion amenable for biopsy or able to provide tissue from biopsy within last 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic, hepatic, and cardiac function

Exclusion Criteria:

* History of allergic reactions to certain components of SBT6050 or similar drugs
* Untreated brain metastases
* Active autoimmune disease or a documented history of autoimmune disease or syndrome
* Human immunodeficiency virus infection, active hepatitis B infection or hepatitis C infection
* Additional protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects experiencing dose limiting toxicities | 28 days
  Part 1 and 3 only
The incidence and severity of adverse events (AEs) and serious adverse events | 2 years
  Parts 1, 2, 3, 4, and 5
Objective response rate, defined as confirmed Complete Response (CR) or Partial Response (PR) | 2 years
  Parts 2, 4, and 5
Duration of response, defined as the time from date of first response (CR or PR) | 2 years
  Parts 2, 4, and 5

SECONDARY OUTCOMES:
Objective response rate, defined as confirmed Complete Response (CR) or Partial Response (PR) | 2 years
  Parts1 and 3 only
Duration of response, defined as the time from date of first response (CR or PR) | 2 years
  Parts 1 and 3 only
Disease control rate, defined as CR, PR, or stable disease for at least 6 months | 2 years
  Parts 1, 2, 3, 4, and 5
Estimates of selected pharmacokinetics (PK ) parameters for SBT6050 | 2 years
  Cmax: Parts 1, 2, 3, 4, and 5
Estimates of selected pharmacokinetics (PK ) parameters for SBT6050 | 2 years
  AUC: Parts 1, 2, 3, 4, and 5
Incidence of antidrug antibodies (ADA) to SBT6050 | 2 years
  Parts 1 and 2
Progression free survival | 2 years
  Parts 2, 4, and 5

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hunder, MD, Study Director — Silverback Therapeutics
Locations (12):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - University of Pittsburgh Medical Center Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute/Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - The START Center for Cancer Care, San Antonio, Texas
- Australia (3):
  - Macquarie University Hospital Clinical Trials Unit, Sydney, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Breast Cancer Research Centre - WA, Nedlands, Western Australia
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No